CLINICAL TRIAL: NCT03416127
Title: Effect of Propolis or Metformin Administration on Glycemic Control in Patients With Type 2 Diabetes Mellitus Without Pharmacological Treatment
Brief Title: Effect of Propolis or Metformin Administration on Glycemic Control in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROPOLIS-METFORMIN-DM2
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus type 2; Glycemic control; Propolis; Metformin; Pharmacological treatment-naïve patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Propolis; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propolis (Experimental): Propolis capsules, 300 mg, two times per day before break-fast and dinner during 12 weeks.
  Interventions: Drug: Propolis
- Metformin (Experimental): Metformin capsules, 850 mg, two times per day before break-fast and dinner during 12 weeks.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo capsules, two times per day before break-fast and dinner during 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propolis — Propolis capsules, 300 mg, two times per day before break-fast and dinner during 12 weeks.
  Arms: Propolis
Drug: Metformin — Metformin capsules, 850 mg, two times per day before break-fast and dinner during 12 weeks.
  Other Names: Metformin hydrochloride
  Arms: Metformin
Drug: Placebo — Calcined magnesium, two times per day before break-fast and dinner during 12 weeks.
  Other Names: Calcined magnesium
  Arms: Placebo

SUMMARY:
The aim of this study was to evaluate the effect of propolis or metformin on glycemic control in patients with type 2 diabetes mellitus without pharmacological treatment.

All patients received for 12 weeks propolis, metformin or placebo. Fasting serum glucose, 2-h serum glucose after oral glucose tolerance test, glycated hemoglobin A1c, a metabolic profile, areas under the curve of glucose and insulin, insulinogenic index, Stumvoll index, and Matsuda index were measured.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial of three pharmacological groups was carried out, with the participation of 36 patients with type 2 Diabetes Mellitus without pharmacological treatment.

At the beginning and end of the study, fasting serum glucose, 2-h serum glucose after oral glucose tolerance test, glycated hemoglobin A1c, and a metabolic profile were measured. Areas under the curve of glucose and insulin, total insulin secretion insulinogenic index), the first phase of insulin secretion (Stumvoll index), and insulin sensitivity (Matsuda index) were calculated.

All patients received for 12 weeks two capsules a day, one before the first bite of breakfast and another before the first bite of dinner. 12 of them took propolis (300 mg), another 12 received metformin (850 mg), and 12 more placebo in the same pharmacological presentation.

This protocol was approved by a local ethics committee and written informed consent was obtained from all volunteers.

Results are presented as mean and standard deviation. Intra-group differences were evaluated using Kruskal-Wallis and Mann-Whitney U-tests, while inter-group differences were calculated with the Wilcoxon test; p≤0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 30 and 60 years
* Mild to moderate physical activity
* Stable body weight for at least 12 weeks prior to the study
* BMI 25.0 - 34.9 kg/m2
* Diabetes mellitus type 2 of recent diagnosis without pharmacological treatment, with one of the following criteria (fasting blood glucose levels >126 mg/dl; or postprandial blood glucose levels after an oral glucose tolerance test with 75 of oral glucose >200 mg/dl
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Previous treatment for glucose
* Fasting glucose ≥250 mg/dL
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Hypersensibility to ingredients of intervention
* Known allergies to bee stings or their derived products
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥240 mg/dL

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — Intstituto de Terapeútica Experimental y Clínica.
Locations (1):
- Intstituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propolis | Metformin | Placebo
Started | 12 | 12 | 12
Completed | 12 | 11 | 11
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propolis | Metformin | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (7) | 51 (4) | 50 (5) | 49 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 7 | 18
  Male | 8 | 5 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 12 | 36
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 12 | 36
Fasting serum glucose [Mean (Standard Deviation); unit: mmol/L] — Fasting serum glucose was analyzed with the glucose oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 7.3 (1.4) | 8.0 (1.6) | 7.7 (1.2) | 7.7 (1.4)
2 hours after OGTT [Mean (Standard Deviation); unit: mmol/L] — 2-h serum glucose was analyzed with the glucose oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 14.6 (2.1) | 15.8 (2.8) | 13.2 (1.9) | 14.5 (2.5)
Glycosylated Hemoglobin (A1C) [Mean (Standard Deviation); unit: percentage] — Glycosylated Hemoglobin (A1C) was evaluated with liquid chromatography method.
  percentage | 6.6 (0.8) | 6.8 (0.9) | 6.8 (0.9) | 6.7 (0.8)
Total insulin secretion [Mean (Standard Deviation); unit: index] — The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔAUC insulin/ΔAUC glucose), the entered values reflect the total insulin secretion
  index | 0.5 (0.1) | 0.4 (0.2) | 0.5 (0.1) | 0.5 (0.1)
Insulin sensitivity [Mean (Standard Deviation); unit: index] — Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
  index | 1.0 (0.4) | 1.1 (0.3) | 0.8 (0.3) | 1.0 (0.3)
First phase of insulin secretion [Mean (Standard Deviation); unit: index] — Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
  index | 2092 (653) | 1608 (736) | 2221 (566) | 1984 (686)
AUC glucose [Mean (Standard Deviation); unit: mmol*min/L] — Area under the curve (AUC) of glucose and insulin was calculated with the polygonal formula.
  mmol*min/L | 965 (137) | 1039 (174) | 930 (90) | 978 (133.6)
AUC insulin [Mean (Standard Deviation); unit: pmol*min/L] — Area under the curve (AUC) of glucose and insulin was calculated with the polygonal formula.
  pmol*min/L | 52541 (9165) | 45323 (9005) | 53869 (5053) | 50577.6 (7741)
Glucose 30 min after oral glucose tolerance test [Mean (Standard Deviation); unit: mmol/L] — Glucose 30' was analyzed with the glucose oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 12.4 (2.3) | 13.7 (3.8) | 12.0 (1.3) | 12.7 (2.7)
Glucose 60 min after oral glucose tolerance test [Mean (Standard Deviation); unit: mmol/L] — Glucose 60' was analyzed with the glucose oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 15.2 (3.0) | 17.2 (2.9) | 14.7 (1.9) | 15.6 (2.7)
Glucose 90 min after oral glucose tolerance test [Mean (Standard Deviation); unit: mmol/L] — Glucose 90' was analyzed with the glucose oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 14.7 (2.0) | 17.5 (2.4) | 14.3 (2.8) | 15.5 (2.8)
Waist circumference [Mean (Standard Deviation); unit: cm] — Waist circumference was measured with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
  cm | 101.2 (9.6) | 103.4 (11.7) | 103.2 (10.2) | 102.6 (10.3)
Body weight [Mean (Standard Deviation); unit: kg] — Body weight was evaluated through a bioimpedance digital scale and results are reported in kg with a decimal.
  kg | 76.4 (11.5) | 80.7 (14.4) | 78.6 (13.1) | 78.6 (12.8)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index was calculated as weight (kg) divided by height (m2).
  kg/m^2 | 29.0 (4.4) | 29.1 (3.7) | 30.2 (3.13) | 29.5 (3.7)
Percentage of fat mass [Mean (Standard Deviation); unit: % fat mass] — Percentage of fat mass was evaluated through bioimpedance.
  % fat mass | 32.8 (9.7) | 30.7 (6.8) | 33.8 (8.3) | 32.4 (8.2)
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] — Total cholesterol was analyzed with the cholesterol oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 5.0 (0.8) | 4.7 (1.1) | 4.7 (0.5) | 4.8 (0.8)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] — Triglycerides were analyzed with the triglycerides oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 2.2 (1.1) | 1.7 (0.6) | 2.0 (1.0) | 2.0 (0.9)
High Density Lipoprotein cholesterol (c-HDL) [Mean (Standard Deviation); unit: mmol/L] — High-density lipoprotein cholesterol (c-HDL) was analyzed with the cholesterol oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 1.0 (0.3) | 0.9 (0.3) | 0.9 (0.2) | 0.9 (0.2)
Low-Density Lipoproteins-cholesterol (c-LDL) [Mean (Standard Deviation); unit: mmol/L] — Low-density lipoprotein-cholesterol (c-LDL) was calculated with the Friedewald formula as follows: LDL-c (mmol/L)= TC (mmol/L) - HDL-c (mmol/L) - [TG(mmol/L)/2.2]
  mmol/L | 3.0 (0.8) | 3.0 (0.8) | 2.9 (0.5) | 3.0 (0.7)
Very low density lipoprotein (VLDL) [Mean (Standard Deviation); unit: mmol/L] — Very low density cholesterol (c-VLDL) was analyzed with the cholesterol oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 1.0 (0.5) | 0.8 (0.3) | 0.9 (0.5) | 0.9 (0.4)
Creatinine [Mean (Standard Deviation); unit: mmol/L] — Creatinine was analyzed with the alkaline picrate technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 72.5 (31.8) | 65.4 (21.2) | 69.8 (27.4) | 70.7 (26.5)
Uric acid [Mean (Standard Deviation); unit: mmol/L] — Uric acid was analyzed with the uric acid oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 356.9 (71.4) | 315.2 (65.4) | 309.2 (89.2) | 327.1 (77.3)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure (SBP) and diastolic (DBP).
  mmHg | 116.9 (8.7) | 118.4 (10.6) | 115.7 (7.2) | 117.0 (8.8)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure (SBP) and diastolic (DBP).
  mmHg | 76.5 (7.8) | 76.2 (7.0) | 73.4 (6.7) | 75.4 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Serum Glucose
Description: The fasting glucose levels were evaluated at week 12 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 12
Time Frame: Week 12
Population: Two of the study groups have one less patient due to withdrawal by subject, as mentioned in the participant flow, so the analysis of this outcome is calculated with those who finished the intervention
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 6.6 (0.9) | 7.3 (1.1) | 8.2 (1.7)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.031, Kruskal-Wallis

2. Primary Outcome: 2 Hours After Oral Glucose Tolerance Test in Week 12
Description: 2-h serum glucose levels were evaluated at week 12 after a oral glucose tolerance test with enzymatic/colorimetric techniques and the entered values reflect the insulin sensitivity at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 13.1 (1.9) | 13.7 (2.7) | 13.2 (2.1)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.963, Kruskal-Wallis

3. Primary Outcome: Glycosylated Hemoglobin (A1C)
Description: Glycosylated hemoglobin was evaluated at week 12 by high pressure liquid chromatography (HPLC) and the entered values reflect the glycosylated hemoglobin at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of A1C
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
% of A1C | 6.3 (0.9) | 6.6 (0.8) | 7.0 (1.0)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.236, Kruskal-Wallis

4. Secondary Outcome: Total Insulin Secretion
Description: Total insulin secretion was calculated at week 12 with insulinogenic index and the entered values reflect the total insulin secretion at week 12.
  The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔAUC insulin/ΔAUC glucose), the entered values reflect the total insulin secretion
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Groups:
- Placebo: Placebo capsules, two times per day before break-fast and dinner during 12 weeks.
  Placebo: Calcined magnesium, two times per day before break-fast and dinner during 12 weeks.
  Period Title: Overall Study
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
index | 0.5 (0.2) | 0.3 (0.2) | 0.5 (0.2)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.015, Kruskal-Wallis

5. Secondary Outcome: Insulin Sensitivity
Description: Insulin sensitivity was calculated at week 12 with Matsuda index and the entered values reflect the insulin sensitivity at week 12.
  Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
index | 1.5 (0.6) | 1.8 (1.0) | 1.0 (0.5)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.017, Kruskal-Wallis

6. Secondary Outcome: First Phase of Insulin Secretion
Description: The first phase of insulin secretion was calculated at week 12 with Stumvoll index and the entered values reflect the frst phase of insulin secretion at week 12.
  Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
index | 1346 (784) | 996 (742) | 1652 (863)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.162, Kruskal-Wallis

7. Secondary Outcome: AUC Glucose
Description: Area under the curve (AUC) of glucose was calculated with the polygonal formula.
  The area under the curve (AUC) of glucose, (0.5 * glucose (G) 0´ + (G 30´+G 60´ + G 90´) + 0.5 * G 120´) * 30; has been widely used for calculating the glycemic index and for evaluating the efficacy of medications for postprandial hyperglycemia.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol*min/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol*min/L | 921 (126) | 967 (116) | 939 (126.4)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.686, Kruskal-Wallis

8. Secondary Outcome: AUC Insulin
Description: Area under the curve (AUC) of insulin was calculated with the polygonal formula.
  The area under the curve (AUC) of insulin, (0.5 * Insulin (I) 0´ + (I 30´+I 60´ + I 90´) + 0.5 * I 120´) * 30; has been widely used for calculating the glycemic index and for evaluating the efficacy of medications for postprandial hyperinsulinemia.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol*min/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
pmol*min/L | 44123 (13381) | 27603 (15935) | 51287 (7440)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.004, Kruskal-Wallis

9. Secondary Outcome: Glucose 30 Min After Oral Glucose Tolerance Test at 12 Week
Description: The glucose levels 30' were evaluated at week 12 with enzymatic/colorimetric techniques and the entered values reflect the glucose 30' at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 12.3 (2.0) | 12.5 (2.1) | 12.0 (1.8)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.945, Kruskal-Wallis

10. Secondary Outcome: Glucose 60 Min After Oral Glucose Tolerance Test at 12 Week
Description: The glucose levels 60' were evaluated at week 12 with enzymatic/colorimetric techniques and the entered values reflect the glucose 60' at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 15.1 (2.8) | 15.9 (2.5) | 14.2 (2.6)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.332, Kruskal-Wallis

11. Secondary Outcome: Glucose 90 Min After Oral Glucose Tolerance Test at 12 Week
Description: The glucose levels 90' were evaluated at week 12 with enzymatic/colorimetric techniques and the entered values reflect the glucose 90' at week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 14.2 (2.6) | 16.6 (2.1) | 14.9 (2.9)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.075, Kruskal-Wallis

12. Secondary Outcome: Waist Circumference
Description: Waist circumference was evaluated at week 12 with a flexible tape
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
cm | 100.7 (10.0) | 102.2 (11.9) | 101.5 (10.2)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.903, Kruskal-Wallis

13. Secondary Outcome: Body Weight
Description: The body weight was measured at week 12 with a bioimpedance balance and the entered values reflect the body weight at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
kg | 75.3 (11.3) | 81.0 (15.2) | 77.8 (13.5)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.697, Kruskal-Wallis

14. Secondary Outcome: Body Mass Index
Description: Body Mas Index was calculated at week 12 with the Quetelet index formula and the entered values reflect the body mass index at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
kg/m2 | 28.6 (4.3) | 29.2 (3.8) | 30.0 (2.9)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.668, Kruskal-Wallis

15. Secondary Outcome: Percentage of Fat Mass
Description: Percentage of fat mass was evaluated through bioimpedance.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of fat mass
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
% of fat mass | 32.8 (10.3) | 28.4 (6.8) | 33.6 (8.2)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.308, Kruskal-Wallis

16. Secondary Outcome: Total Cholesterol
Description: Total cholesterol levels were evaluated at week 12 by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 5.1 (0.7) | 4.6 (0.9) | 4.7 (0.7)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.318, Kruskal-Wallis

17. Secondary Outcome: Triglycerides
Description: Triglycerides levels were evaluated at week 12 with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 2.0 (0.8) | 2.0 (1.0) | 1.9 (0.8)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.880, Kruskal-Wallis

18. Secondary Outcome: High Density Lipoprotein Cholesterol (c-HDL)
Description: c-HDL levels were evaluated at week 12 with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 1.0 (0.3) | 0.9 (0.2) | 0.9 (0.1)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.376, Kruskal-Wallis

19. Secondary Outcome: Low Density Lipoproteins Cholesterol (c-LDL)
Description: c-LDL levels were evaluated at week 12 with enzymatic/colorimetric techniques and the entered values reflect the c-LDL level at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 3.1 (0.5) | 2.7 (0.5) | 3.0 (0.5)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.210, Kruskal-Wallis

20. Secondary Outcome: Very Low Density Lipoprotein (c-VLDL)
Description: Very low density lipoprotein (c-VLDL) was analyzed with the cholesterol oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 0.9 (0.4) | 0.9 (0.5) | 0.9 (0.4)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.880, Kruskal-Wallis

21. Secondary Outcome: Creatinine
Description: Creatinine levels were evaluated at week 12 with enzymatic/colorimetric techniques
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 55.7 (10.6) | 74.2 (16.8) | 63.6 (26.5)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.059, Kruskal-Wallis

22. Secondary Outcome: Uric Acid
Description: Uric acid levels were evaluated at week 12 with enzymatic/colorimetric techniques
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmol/L | 339.0 (77.3) | 327.1 (71.4) | 333.1 (95.2)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.978, Kruskal-Wallis

23. Secondary Outcome: Systolic Blood Pressure
Description: The systolic blood pressure was evaluated at week 12 with a digital sphygmomanometer and the entered values reflect the systolic blood pressure at week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmHg | 114.6 (7.4) | 119.2 (11.4) | 112.8 (6.4)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.122, Kruskal-Wallis

24. Secondary Outcome: Diastolic Blood Pressure
Description: The diastolic blood pressure was evaluated at week 12 with a digital sphygmomanometer and the entered values reflect the diastolic blood pressure at week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | Propolis | Metformin | Placebo
Number analyzed (Participants) | 12 | 11 | 11
mmHg | 74.8 (7.4) | 74.4 (7.9) | 72.3 (3.8)
Statistical Analysis 1: Comparison: Propolis vs Metformin vs Placebo; Test type: Other; p = 0.551, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Throughout the study, an average of 12 weeks
Arm/Group | Propolis | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 3/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propolis (N=12) | Metformin (N=12) | Placebo (N=12)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Loose stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03416127/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03416127/ICF_001.pdf